CLINICAL TRIAL: NCT05720936
Title: A Multicenter Observational Study on In-hospital Stellate Ganglion Block for Arrhythmic Storm
Brief Title: In-hospital Stellate Ganglion Block for Arrhythmic Storm
Acronym: STAR
Status: Recruiting | Type: Observational
Sponsor: Fondazione IRCCS Policlinico San Matteo di Pavia (Other)
Responsible Party: Principal Investigator, Simone Savastano, Principal Investigator, Fondazione IRCCS Policlinico San Matteo di Pavia
Other Study IDs: STAR Study
Record Dates: First submitted 2023-01-07; First posted 2023-02-09 (Actual); Last update posted 2025-06-08 (Actual); Status verified 2025-06

CONDITIONS: Arrhythmic Storm; Electrical Storm; Ventricular Fibrillation; Ventricular Tachycardia
Keywords: PSGB; L-PSGB; Percutaneous Stellate Ganglion Block; Percutaneous Stellate Ganglion Blockade; Electrical Storm
MeSH Terms: conditions — Ventricular Fibrillation; Tachycardia, Ventricular

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- patients with electric storm: patients with electric storm defined as the occurrence of at least three episodes of ventricular fibrillation/tachycardia in 24 hours
  Interventions: Procedure: Percutaneous stellate ganglion block (PSGB)

INTERVENTIONS:
Procedure: Percutaneous stellate ganglion block (PSGB) — Both the two approaches present in literature and commonly used for this technique are allowed for the study:
  * The "anatomical" approach which consist in the identification of the Chassaignac's tubercle that represents the point of needle insertion
  * The "echo-guided" approach

SUMMARY:
Arrhythmic storm is a real emergency and its treatment could be challenging. Antiarrhythmic drugs are few and often ineffective. Neuromodulation has been grown in evidences but no large multicentric studies are present in literature about safety and effectiveness of Percutaneous Stellate Ganglion Block (PSGB). Patients with an electrical storm refractory to at least one antiarrhythmic drug will receive PSGB and will be enrolled in the present study.

The number of defibrillations before and after the treatment will be compared, complications will be annotated.

DETAILED DESCRIPTION:
This is an international multicenter observational retrospective and prospective short term (24 hours) longitudinal study, promoted and coordinated by the Fondazione IRCCS Policlinico San Matteo of Pavia (Italy).

Materials and methods:

All the patients who will meet the inclusion criteria will be enrolled in the study. Conscious patients with a sufficient free interval between arrhythmic relapses will sign the informed consent for the procedure and for data collection (attached at the study protocol) before the procedure. In case of unconscious patients the medical doctor will perform the procedure being in an emergency situation and the inform consent for data collection will be signed afterward once possible.

Inclusion criteria:

All the patients presenting with an arrhythmic storm defined as more than three sustained ventricular arrhythmias in 24 hours refractory to the standard medical treatment.

Exclusion criteria:

* A previous history of cardiac sympathicectomy
* Having a neck judged by the doctor as non-suitable for the procedure (previous neck surgery, previous burns, presence of large scars, thyroid goiter)

PSGB technique:

Both the two approaches present in literature and commonly used for this technique are allowed for the study:

* The "anatomical" approach which consist in the identification of the Chassaignac's tubercle that represents the point of needle insertion
* The "echo-guided" approach Regardless to the approach (anatomical or echo-guided) the doctor will be able to choose, according to the clinical characteristics of the patients, whether to perform a single shot injection of anesthetic or a continuous infusion of anesthetic. In the second case a catheter will be left in place and connected to an infusion pump.

Study Objectives:

The primary objective is the effectiveness of the PSGB expressed by the reduction of arrhythmic relapses [number of Direct Current (DC) shocks or Anti-Tachycardia Pacing ATP] in the 12 hours immediately after the PSGB as compared to the 6 hours immediately preceding the PSGB of at least 50%.

The secondary objectives are:

1. The comparison of the number of shocks 12h before and 12h after the procedure
2. The feasibility of the procedure expressed as the number of complications within 12 hours from the procedure. The following complications will be considered:

   * Simple hematoma
   * Symptoms due to anesthetic absorbance
   * Hematoma requiring intervention
   * Intravascular injection without complication
   * Intravascular injection with complication
   * Brachial plexus damage
   * Simple vascular damage
   * Vascular damage requiring intervention
3. The comparison of the effectiveness endpoint in patients with and without the appearance of anisocoria
4. The comparison of effectiveness between patients who will receive "anatomical" PSGB and those who will receive echo-guided PSGB
5. The comparison of effectiveness between patients who will receive anaesthetic infusion in the site of PSGB as compared to those who will not.

Statistics:

Sample size: The investigators plan to enroll patients satisfying the inclusion/exclusion criteria over a time horizon of 5 years. Based on our previous experience over the previous 18 months (enrollment of 8 patients) about 5 patients per year are though to be enrolled, thus reaching a sample size 33 patients in the Pavia Center. The success is effectiveness to be not less then 90%, based on our historical cohort. This will yield a confidence interval of 76% to 98%, corresponding to a precision of 11%. Also, with this sample size it will be able to exclude an effectiveness of 70% (considered as the lower bound of acceptability) with a power of 94% (alpha 2-sided 5%).

With the inclusion of further centers, the increased sample size will allow an increased precision of the estimates; for instance for 100 patients precision would be 6.5% (first step already achieved) and for 500 patients would be 2.6%.

Statistical analysis: Data will be described with the mean and standard deviation or the median and 25th-75th percentile if continuous and counts and percent if categorical.

For the analysis of the primary endpoint the rate of effectiveness together with its 95% exact binomial confidence interval will be computed.

Data management:

Data will be collected using the REDCap platform (e-CRF). A personal and password protected account will be created for each investigator who will be able to access only to the data from his/her Center.

ELIGIBILITY:
Inclusion Criteria:

* age ≥ 18 years,
* presence of arrhythmic storm defined as more than three sustained ventricular arrhythmias in 24 hours refractory to the standard medical treatment.

Exclusion Criteria:

* A previous history of cardiac sympathicectomy
* Having a neck judged unsuitable for the procedure (previous neck surgery, previous burns, presence of large scars, thyroid goiter)

Both the two approaches present in literature and commonly used for this technique are allowed for the study:

* The "anatomical" approach which consist in the identification of the Chassaignac's tubercle that represents the point of needle insertion
* The "echo-guided" approach Regardless to the approach (anatomical or echo-guided) the doctor will be able to choose, according to the clinical characteristics of the patients, whether to perform a single shot injection of anesthetic or a continuous infusion of anesthetic. In the second case a catheter will be left in place and connected to an infusion pump.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All the patients who will meet the inclusion criteria will be enrolled in the study. Conscious patients with a sufficient free interval between arrhythmic relapses will sign the informed consent for the procedure and for data collection (attached at the study protocol) before the procedure. In case of unconscious patients the medical doctor will perform the procedure being in an emergency situation and the inform consent for data collection will be signed afterward once possible.
Sampling Method: Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2017-11-07 (Actual); Primary Completion 2028-12-31 (Estimated); Study Completion 2028-12-31 (Estimated)

PRIMARY OUTCOMES:
reduction of arrhythmic relapses after PSGB | 12h before and 12h after the procedure
  effectiveness of the PSGB expressed by the reduction of arrhythmic relapses (number of DC shocks or anti-tachycardia pacing ATP) of at least 50% after PSGB.

SECONDARY OUTCOMES:
reduction of arrhythmic relapses after PSGB | 12h before and 12h after the procedure
  the effectiveness of the technique will be evaluated by the comparison of the number of shocks before and after the procedure
complication rate related to PSGB | 12 hours after the procedure
  The feasibility of the procedure will be expressed as the number of complications within 12 hours from the procedure. The following complications will be considered:
  * Simple hematoma
  * Symptoms due to anesthetic absorbance
  * Hematoma requiring intervention
  * Intravascular injection without complication
  * Intravascular injection with complication
  * Brachial plexus damage
  * Simple vascular damage
  * Vascular damage requiring intervention
relationship between the appearance of anisocoria and the reduction of arrhythmic relapses after PSGB | 12h before and 12h after the procedure
  The comparison of the effectiveness endpoint in patients with and without the appearance of anisocoria
relationship between the approach used and the reduction of arrhythmic relapses after PSGB | 12h before and 12h after the procedure
  The comparison of effectiveness between patients who will receive "anatomical" PSGB and those who will receive echo-guided PSGB.
relationship between the administration type and the reduction of the arrhythmic relapses after PSGB. | 12h before and 12h after the procedure
  The comparison of effectiveness between patients who will receive continuous anesthetic infusion and patients who will receive a single bolus in the site of PSGB.

CONTACTS AND LOCATIONS:
Locations (38):
- Italy (37):
  - A.O. SS. Antonio e Biagio e Cesare Arrigo di Alessandria., Alessandria, AL
  - Ospedale di Bentivoglio, Bentivoglio, BO
  - Ospedale Maggiore di Bologna, Bologna, BO
  - Cardiology Department, Fondazione IRCCS Policlinico San Matteo, Pavia, PV
  - Ospedale Civile, Voghera, PV
  - Ospedale Mater Salutis, Legnago, VR
  - A.O.U. delle Marche, Ospedali Riuniti, Ancona
  - Ospedale Cardinal Massaia, Asti
  - Policlinico S. Orsola-Malpighi, IRCCS A.O.U. Bologna, Bologna
  - P.O. "San Michele" dell'ARNAS "G. Brotzu" di Cagliari, Cagliari
  - Istituto clinico Humanitas Mater Domini di Castellanza, Castellanza
  - Ospedale Maggiore, Crema
  - Ospedale San Biagio di Domodossola, Domodossola
  - Ospedale S. Maria Annunziata, Florence
  - P.O. Santa Maria Nuova e Palagi, Florence
  - Ospedale Misericordia di Grosseto., Grosseto
  - Ospedale di Gubbio-Gualdo Tadino, USL Umbria 1, Gubbio
  - Ospedale Civile di Ivrea, Ivrea
  - Ospedale Alessandro Manzoni, Lecco
  - Azienda USL Toscana Nord Ovest, Presidio di Livorno, Livorno
  - A.O.U. Policlinico "G. Martino" di Messina., Messina
  - ASST Santi Paolo e Carlo, Milan
  - IRCCS Ospedale San Raffaele, Milan
  - Istituto Auxologico Italiano, Milan
  - ASST Grande Ospedale Metropolitano Niguarda di Milano, Milan
  - Ospedale V. Monaldi - AOS dei Colli, Napoli
  - A.O.U. Maggiore della Carità di Novara, Novara
  - Azienda Ospedale Università Padova, Padua
  - Ospedale S. Maria della Misericordia - Perugia, Perugia
  - Ospedale "Infermi" AUSL Romagna, Rimini
  - A.O.U. Ospedale Sant'Andrea, Roma
  - Fondazione Policlinico Universitario Agostino Gemelli, Università Cattolica del Sacro Cuore, Roma
  - Fondazione PTV Policlinico Tor Vergata di Roma, Roma
  - Ospedale Fatebenefratelli di Roma., Roma
  - Ospedale San Paolo, Savona
  - Ospedale Molinette di Torino, Torino
  - Azienda Ospedaliera Universitaria Integrata - Verona, Verona
- Istituto Cardiocentro Ticino, Lugano, Switzerland

IPD SHARING:
Plan to Share IPD: Undecided
every study site will be able to have data regarding their patients

REFERENCES:
- [Background] Savastano S, Schwartz PJ. Blocking nerves and saving lives: Left stellate ganglion block for electrical storms. Heart Rhythm. 2023 Jul;20(7):1039-1047. doi: 10.1016/j.hrthm.2022.11.025. Epub 2022 Dec 9. PMID 36509320
- [Background] Savastano S, Dusi V, Baldi E, Rordorf R, Sanzo A, Camporotondo R, Fracchia R, Compagnoni S, Frigerio L, Oltrona Visconti L, De Ferrari GM. Anatomical-based percutaneous left stellate ganglion block in patients with drug-refractory electrical storm and structural heart disease: a single-centre case series. Europace. 2021 Apr 6;23(4):581-586. doi: 10.1093/europace/euaa319. PMID 33190159
- [Background] Savastano S, Pugliese L, Baldi E, Dusi V, Tavazzi G, De Ferrari GM. Percutaneous continuous left stellate ganglion block as an effective bridge to bilateral cardiac sympathetic denervation. Europace. 2020 Apr 1;22(4):606. doi: 10.1093/europace/euaa007. No abstract available. PMID 32034906
- [Background] Savastano S, Baldi E, Camporotondo R, Belliato M, Marinoni B, De Ferrari GM. Percutaneous stellate ganglion block and extracorporeal cardiopulmonary resuscitation: an effective and safe combination for refractory ventricular fibrillation. Europace. 2020 Jan 1;22(1):148. doi: 10.1093/europace/euz180. No abstract available. PMID 31257420
- [Background] Zeppenfeld K, Tfelt-Hansen J, de Riva M, Winkel BG, Behr ER, Blom NA, Charron P, Corrado D, Dagres N, de Chillou C, Eckardt L, Friede T, Haugaa KH, Hocini M, Lambiase PD, Marijon E, Merino JL, Peichl P, Priori SG, Reichlin T, Schulz-Menger J, Sticherling C, Tzeis S, Verstrael A, Volterrani M; ESC Scientific Document Group. 2022 ESC Guidelines for the management of patients with ventricular arrhythmias and the prevention of sudden cardiac death. Eur Heart J. 2022 Oct 21;43(40):3997-4126. doi: 10.1093/eurheartj/ehac262. No abstract available. PMID 36017572